CLINICAL TRIAL: NCT06827704
Title: Physical Activity Targeting Metabolic Syndrome for Prevention of Breast Cancer in South Asian Indian Immigrant Women
Brief Title: Physical Activity Targeting Metabolic Syndrome for Prevention of Breast Cancer in SAI Women
Acronym: MetS-BC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 24032906-IRB01; DUNS: 068610245 (Other: Rush University Medical Center)
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Metabolic Syndrome; Breast Cancer Prevention; Physical Activity
MeSH Terms: conditions — Metabolic Syndrome; Motor Activity

STUDY DESIGN:
Intervention Model Description: 2x2 factorial design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Enhanced physical activity monitor which is Fitbit watch with mobile App (Experimental): Participants will receive an enhanced physical activity monitor treatment for 6 months which includes goal setting with a physical activity prescription, and self-monitoring with a physical activity monitor (Fitbit watch).
  Interventions: Behavioral: Enhanced physical activity monitor which is Fitbit watch with mobile App
- Bollywood-style group dance (Experimental): Participants will participate in 60-minute, moderate-intensity Bollywood-style culturally tailored group dance virtual sessions, 2x/week for 6 months.
  Interventions: Behavioral: Bollywood-style group dance
- PAMDance (Experimental): Participants will receive an enhanced physical activity monitor treatment for 6 months which includes goal setting with a physical activity prescription, and self-monitoring with a physical activity monitor (Fitbit watch). In addition, Participants will participate in 60-minute, moderate-intensity Bollywood-style culturally tailored group dance virtual sessions, 2x/week for 6 months.
  Interventions: Behavioral: PAMDance
- Usual care control (No Intervention): Participants in the usual care group do not receive any PAM or Dance related intervention.

INTERVENTIONS:
Behavioral: Enhanced physical activity monitor which is Fitbit watch with mobile App — Participants will receive an enhanced physical activity monitor treatment for 6 months which includes goal setting with a physical activity prescription, and self-monitoring with a physical activity monitor (Fitbit watch). Edit
  Arms: Enhanced physical activity monitor which is Fitbit watch with mobile App
Behavioral: Bollywood-style group dance — Participants will participate in 60-minute, moderate-intensity Bollywood-style culturally tailored group dance virtual sessions, 2x/week for 6 months
  Arms: Bollywood-style group dance
Behavioral: PAMDance — Participants will receive an enhanced physical activity monitor treatment for 6 months which includes goal setting with a physical activity prescription, and self-monitoring with a physical activity monitor (Fitbit watch). In addition, Participants will participate in 60-minute, moderate-intensity Bollywood-style culturally tailored group dance virtual sessions, 2x/week for 6 months
  Arms: PAMDance

SUMMARY:
This study aims to to improve physical activity and metabolic outcomes for breast cancer prevention in South Asian Indian immigrant women.

DETAILED DESCRIPTION:
One out of every eight SAI women in the US is at risk of developing breast cancer and breast cancer manifests 5-10 years earlier in South Asian Indian immigrant (SAI) women (54.5 [SD =13.3]) than in their non-Hispanic White women counterparts (p<.01). The risk of breast cancer is 2.3 times higher in SAI women with metabolic syndrome (hypertension, insulin resistance, dyslipidemia, and central obesity (HR 2.30, 95% CI 1.18-4.49) than their non-Hispanic White women counterparts. To reduce disparities related to metabolic syndrome associated breast cancer in at-risk SAI women, increasing lifestyle physical activity is critical. Approximately 50% of first-generation SAI women in the US, fail to meet recommended physical activity guidelines. Western leisure-time activities lack the cultural connection for many SAI women due to language issue, perceived racial discrimination, and a limited sense of community. To address disparities related to physical activity barriers, the physical activity interventions must be culturally tailored to promote their uptake among at-risk first-generation midlife SAI women. In-person culturally tailored program with Bollywood-style group dance and goal setting with a physical activity monitor have been shown to significantly improve average daily steps, self-efficacy, blood pressure, blood glucose, lipids, body weight, and waist circumference (p<.05) in first-generation midlife SAI women. However, lack of time due to role expectations at home and lack of transportation presented a challenge for SAI women to attend in-person behavioral group activities. Therefore, the purpose of this virtual 24-week culturally relevant physical activity program with 2x2 factorial design is to improve physical activity and metabolic outcomes for breast cancer prevention in first-generation midlife (aged 40-65) SAI women with insufficient physical activity (self-reported <150 minutes/week of moderate-intensity or <75 minutes/week of vigorous-intensity physical activity in the past month). Women (N=96) will be randomized into one of four conditions 1) Enhanced physical activity monitor which is Fitbit watch with mobile App (PAM), 2) Bollywood-style group dance (Dance), 3) PAMDance, or 4) usual care control. This study aims to: (1) Determine the independent and combined efficacies of PAM and Dance at 12 and 24 weeks on lifestyle physical activity (steps/day [ActiGraph], minutes of moderate to vigorous physical activity/week (ActiGraph and self-report) in midlife SAI women; (2) Determine the independent and combined efficacies of PAM and Dance at 12 and 24 weeks on metabolic outcomes (blood pressure, blood glucose, lipids, body mass index, and waist circumference). We expect that our findings will demonstrate the efficacy of a virtual culturally tailored lifestyle behavioral physical activity intervention to be broadly applicable for addressing metabolic disparities that confer increased risk for breast cancer in first-generation midlife SAI women.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified first-generation SAI woman aged 40-65 years without breast cancer diagnosis (permanent residency in US or are in the process of obtaining permanent residency)
* Insufficiently active (self-reported <150 minutes/week of moderate-intensity or <75 minutes/week of vigorous-intensity PA in the past month)
* Conversant in Hindi
* Owns a smartphone for Fitbit application
* Has a computer or mobile device with Internet access
* Willing to participate in recorded Virtual intervention sessions
* Medical clearance if has Type 1 diabetes, or Type 2 diabetes with an A1C ≥ 9.0%, or have an A1C of ≥ 6.5% without a prior diabetes diagnosis
* Has no disabilities preventing regular PA determined by Physical Activity Readiness Questionnaire (PAR-Q & You)

Exclusion Criteria:

* Major signs/symptoms of pulmonary or CVD, unstable cardiac or pulmonary disease in the past month, or other conditions interfering with walking (per PAR-Q & You)
* Systolic BP ≥160 and/or diastolic BP ≥100

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identified first-generation South Asian Indian immigrant woman
Enrollment: 96 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical Activity- Steps/day | Baseline plus change will be assessed at weeks 12 and 24.
  Determine the independent and combined efficacies of PAM and Dance at 12 and 24 weeks on lifestyle PA (steps/day [ActiGraph] in midlife SAI women.
Physical Activity- Moderate to Vigorous Physical Activity (MVPA)/day | Baseline plus change will be assessed at weeks 12 and 24.
  Determine the independent and combined efficacies of PAM and Dance at 12 and 24 weeks on minutes of Moderate to Vigorous Physical Activity (MVPA)/day (ActiGraph and self-report) in midlife SAI women.

SECONDARY OUTCOMES:
Metabolic outcomes (1) | Baseline plus change will be assessed at weeks 12 and 24.
  Blood pressure
Metabolic outcomes (2) | Baseline plus change will be assessed at weeks 12 and 24.
  Blood glucose: point-of-care HbA1C
Metabolic outcomes (3) | Baseline plus change will be assessed at weeks 12 and 24.
  Lipid panel : point-of-care total cholesterol, triglycerides, HDL, LDL
Metabolic outcomes (4) | Baseline plus change will be assessed at weeks 12 and 24.
  Body composition: BMI (weight measured in pounds; height measured in inches)
Metabolic outcomes (5) | Baseline plus change will be assessed at weeks 12 and 24.
  Body composition: waist measured in inches

CONTACTS AND LOCATIONS:
Overall Officials: Manju Daniel, PhD, Principal Investigator — Rush University College of Nursing
Locations (2):
- United States (2):
  - Rush University College of Nursing, Chicago, Illinois
  - Rush University College of Nursing, Sugar Grove, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Daniel M, Miller A, Wilbur J. Multiple instrument translation for use with South Asian Indian immigrants. Res Nurs Health. 2011 Oct;34(5):419-32. doi: 10.1002/nur.20450. Epub 2011 Aug 4. PMID 21818758
- [Background] Daniel M, Abendroth M, Erlen JA. Barriers and Motives to PA in South Asian Indian Immigrant Women. West J Nurs Res. 2018 Sep;40(9):1339-1356. doi: 10.1177/0193945917697218. Epub 2017 Mar 10. PMID 28281387
- [Background] Daniel M, Marquez D, Ingram D, Fogg L. Group Dance and Motivational Coaching for Walking: A Physical Activity Program for South Asian Indian Immigrant Women Residing in the United States. J Phys Act Health. 2021 Mar 1;18(3):262-271. doi: 10.1123/jpah.2019-0316. Epub 2021 Feb 4. PMID 33540381
- [Background] Daniel M, Wilbur J, Fogg LF, Miller AM. Correlates of lifestyle: physical activity among South Asian Indian immigrants. J Community Health Nurs. 2013;30(4):185-200. doi: 10.1080/07370016.2013.838482. PMID 24219639
- [Background] Daniel M, Wilbur J, Marquez D, Farran C. Lifestyle physical activity behavior among South Asian Indian immigrants. J Immigr Minor Health. 2013 Dec;15(6):1082-9. doi: 10.1007/s10903-013-9842-4. PMID 23686529
- [Background] Daniel M, Wilbur J. Physical activity among South Asian Indian immigrants: an integrative review. Public Health Nurs. 2011 Sep-Oct;28(5):389-401. doi: 10.1111/j.1525-1446.2010.00932.x. Epub 2011 May 9. PMID 22092422
- [Background] Daniel M, Buchholz S, Fogg L. Physical Activity in South Asian Indians: A Systematic Review of Randomized Controlled Trials. West J Nurs Res. 2023 Apr;45(4):363-374. doi: 10.1177/01939459221134373. Epub 2022 Nov 2. PMID 36324264